CLINICAL TRIAL: NCT01273649
Title: Therapeutic Effects of Cryotherapy and Transcutaneous Nerves Stimulation on Arthrogenic Muscle Inhibition in Patients With Anterior Cruciate Ligament Reconstruction
Brief Title: Therapeutic Effects of Cryotherapy on Arthrogenic Muscle Inhibition in Patients With Cruciate Ligament Reconstruction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201007065R
Record Dates: First submitted 2011-01-06; First posted 2011-01-10 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Anterior Cruciate Ligament Injury
Keywords: muscle activation; ACL reconstruction; cryotherapy; TENS
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ice, rate of force development (Experimental): to monitor the long term effect of cryotherapy in rate of force development.
  Interventions: Device: cryotherapy

INTERVENTIONS:
Device: cryotherapy — cryotherapy is given with other physical training

SUMMARY:
Anterior cruciate ligament(ACL) injury is one of the most common sport injuries. The major problem after ACL reconstruction or rehabilitation program is quadriceps weakness. Previous studies suggested that cryotherapy and transcutaneous electrical nerve stimulation(TENS) can effectively reduce the arthrogenic muscle inhibition caused by experimental swelling.

Objective:

To exam the effects of 12 weeks cryotherapy and TENS on arthrogenic muscle inhibition in subjects with ACL reconstruction.

Design:

Prospective study.

Subjects:

Male subjects with isolated ACL injury, age between 18~40 years old are going to receive an ACL reconstruction surgery.

Methods:

Quadriceps activation level, quadriceps peak torque during maximal voluntary contraction and rate of force development are measure at presurgery, 3-month, 6-month after surgery. After surgery, subjects will receive 12 weeks, 3 days/week, training programs included 20 minutes cryotherapy and exercise training with TENS.

Data analysis:

Data will be analyzed using SPSS 13.0 software (SPSS Inc., Chicago, IL). One-way ANOVA will be used to analysis data.

DETAILED DESCRIPTION:
Examination procedure:

1. Skin preparation and EMG setting.
2. Fill out knee joint function questionnaire.
3. Warmup with a stationary bike.
4. Single hop for distance.
5. MVIC test and EMG recording.
6. Endurance test.
7. Record surface EMG of vastus lateralis, vastus medialis, biceps femoris and semitendinosus during maximal voluntary contraction.

ELIGIBILITY:
Inclusion Criteria:

* Male subjects with isolated ACL injury, age between 18~40 years old are going to receive an ACL reconstruction surgery.

Exclusion Criteria:

* meniscus lesion, bony fracture and osteochondral lesions

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-09 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Muscle activation | 6 months
  To provide information of individual muscles for the correlation analyses, parameters of muscle activation, such as the integrated electromyography (EMG) normalized to the maximal M wave, are favored.

CONTACTS AND LOCATIONS:
Overall Officials: HK Wang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University, Taipei, Taiwan, Taiwan